CLINICAL TRIAL: NCT03535402
Title: Measurement of the Structural Efficacy in Active Rheumatoid Arthritis (RA) Patients Treated With Sarilumab in Combination With Methotrexate (MTX) and Naive to Biologics as Measured by Low-field MRI Using a Modified OMERACT-RAMRIS Score.
Brief Title: Measurement of the Structural Efficacy in Active RA Patients Treated With Sarilumab in Combination With MTX and Naive to Biologics
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gaylis, Norman B., M.D. (Individual)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RA-012018
Record Dates: First submitted 2018-05-09; First posted 2018-05-24 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — sarilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- open label treatment (Other): single arm with patients receiving 200 mg SC twice a week of sarilumab
  Interventions: Drug: Sarilumab

INTERVENTIONS:
Drug: Sarilumab — SC administration of 200 mg twice a week

SUMMARY:
This is a single site study to determine the structural efficacy of sarilumab when administered to biologic naive patients with active rheumatoid arthritis

DETAILED DESCRIPTION:
This is a single site Phase III 48-week open-label study to evaluate the structural response of sarilumab 200 mg SC injection administered to active RA patients. Active RA is defined as having a Clinical Disease Activity Index (CDAI) >10.0. All patients will have had an inadequate response to MTX (treated with 12.5-20 mg/wk. for at least 3 months) and have had no prior exposure to biologic medications for RA. The MTX will be continued throughout the trial allowing for dose reduction at the Primary Investigator's discretion due to safety. There will be a total of twenty (20) patients enrolled into the trial.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patient must be at least 18 years old at the screening visit. 2. Patient must be able to understand the information provided to them and to give written Informed Consent before any study-related procedures are performed.

  3. Female patients must be either postmenopausal for at least 1 year, surgically incapable of childbearing, or effectively practicing an acceptable method of contraception (oral/parenteral/implantable hormonal contraceptives, IUD, or barrier and spermicide). Abstinence only is not an acceptable method. Patients must agree to use adequate contraception during the study and for 4 weeks after their last dose of sarilumab. Male patients must agree to ensure they or their female partner(s) are using adequate contraception during the study and for 4 weeks after the patient receives their last dose of sarilumab.

  4. Patients must have a diagnosis of adult-onset RA according to the ACR/EULAR (2010) Rheumatoid Arthritis Classification Criteria.

  5. Patients must be experiencing moderate to severe RA, have at least 4 tender and 4 swollen joints at screening and a CDAI score of >10.0 despite treatment with MTX 12.5-20 mg/wk.

  6. Continuous treatment with MTX (12.5-20 mg/wk. orally or intramuscular) for at least 12 weeks prior to screening with a stable dose for the past 4 weeks.

  7. A Baseline MRI must show the presence of osteitis, synovitis or erosions in the hand or wrist.

  8. Patients must be able and willing to comply with the requirements of the study protocol.

Exclusion Criteria:

* 1. Patients who have a diagnosis of any other inflammatory arthritis (e.g., psoriatic arthritis or ankylosing spondylitis) 2. Patients with exposure to biologic medications for RA 3. Patients with a non-inflammatory type of arthritis (e.g. osteoarthritis or fibromyalgia) that in the Investigator's opinion is symptomatic enough to interfere with evaluation of the effect of study drug on the patient's primary diagnosis of RA 4. Patients with history of an infected joint prosthesis at any time with that prosthesis still in situ 5. Patients who are not candidates for treatment with sarilumab as defined by the US Package Insert.

  1. NSAIDs /COX-2 inhibitors any change in treatment or dose-adjustment within 2 weeks prior to screening
  2. Oral corticosteroids >10 mg daily within 4 weeks of baseline
  3. IM/IV/IA corticosteroids any dose 28 days prior to baseline 6. Female patients who are breast-feeding, pregnant, or plan to become pregnant during the trial or within twelve weeks following last dose of study drug 7. Patients with a history of chronic infection due to fungal, parasitic or mycotic pathogens during the preceding year, recent serious or life-threatening infection within 6 months (including herpes zoster), or any current sign or symptom that may indicate an infection 8. Patients with active TB (or history of active TB), positive chest X-ray for TB, or positive (defined as induration of ≥ 5mm) PPD skin test, positive QuantiFERON, or patients having close contact with an individual with active TB. Patients having a PPD skin test ≥ 5 mm or a positive QuantiFERON test can enter the study, provided that active TB is excluded by chest x-Ray and provided that they are adequately treated for latent TB (INH therapy) for 9 months and provided that appropriate treatment is initiated simultaneously with the first administration of sarilumab 9 Patients at a high risk of infection (e.g. leg ulcers, indwelling urinary catheter and persistent or recurrent chest infections and patients who are permanently bedridden or wheelchair bound) 10. Patients with a known allergy or intolerance to sarilumab 11. Prior or current history of malignancy, including lymphoproliferative diseases, other than adequately treated carcinoma in-situ of the cervix, nonmetastatic squamous cell or basal cell carcinoma of the skin, within 5 years prior to randomization (baseline) visit 12. Patients with a current or recent history of severe, progressive, and/or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurological or cerebral disease 13. Patients with class III or IV congestive heart failure according to the New York Heart Association (NYHA) 1964 classification criteria 14. Patients with a history of, or suspected, demyelinating disease of the central nervous system (e.g. multiple sclerosis or optic neuritis) 15. Patients with any other condition (e.g. clinically significant laboratory values) which in the Investigator's judgment would make the patient unsuitable for inclusion in the study 16. Patients who have a metal device affected by MRI (e.g., any type of electronic, mechanical, or magnetic implant; cardiac pacemaker; aneurysm clip(s); implanted cardioverter defibrillator; or a cochlear implant) 17. Patients who have a potential ferromagnetic foreign body (metal slivers, metal shavings, other metal objects) for which they have sought medical attention 18. Concurrent steroid use > 10 mg daily for any concomitant disease 19. Subjects who are known to be HIV, Hepatitis B or Hepatitis C positive 20. Any patient who has surgery within 4 weeks prior to screening or with planned surgery during the course of the study 21. Patients with a history of inflammatory bowel disease or severe diverticulitis or previous gastrointestinal perforation 22. Patients with any of the following laboratory abnormalities at the screening visit:

     * Hemoglobin < 9.0 g/dL
     * White blood cells (WBC) <3000/mm3
     * Neutrophils < 2.0/mm3
     * Platelet Count <150,000/mm3
     * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 1.5 ULN unless documented Gilbert's disease diagnosed by genetic testing
     * Presence of severe uncontrolled hypercholesterolemia (>350 mg/dL) or hyper-
     * triglyceridemia (>500 mg/dL)
     * Bilirubin > ULN unless documented Gilbert's disease diagnosed by genetic testing 23. Prior treatment with sarilumab 24. Treatment with any live or attenuated vaccine within 3 months prior to the Randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Structural Efficacy of Sarilumab | 48 week
  To explore the structural efficacy of sarilumab on synovitis, osteitis, and joint erosions as measured by MRI in active RA patients who had an inadequate response to MTX using the change in the OMERACT RAMRIS score from Baseline to Week 48. Synovitis is graded 0-3 (normal, mild, moderate and severe) as estimated by thirds of the presumed maximum volume of enhancing tissue. Bone edema is graded by percentage volume (0-3),byt 33% volume increments) of the assessed bone. Bone erosion is graded by assessing percentage volume (1-10,by 10 % volume increments) of the assessed bone volume. There are multiple parameters for these measurements and the OMERACTguide has to be used to perform this analysis.

SECONDARY OUTCOMES:
Clinical Response | 48 weeks
  To explore the clinical response of these patients from Baseline to Week 48 as measured by the Clinical Disease Activity Index (CDAI) score. CDAI =28 Swollen Joint Count+28 Tender Joint Count+Provider Global Assessment +Patient Global Assessment. Result Intrepretaion is Remission is <2.8 or equal to 2.8; Low Disease Activity is >2.8 to 10.0; Moderate Disease Activity is 10.0; High Disease Activity is >10.0 to 22.0
Compare Clinical and Structural Efficacy | 48 weeks
  To compare the clinical using the CDAI score and structural outcomes using the Modified OMERACT-RAMRIS score at Week 48 and see if there is a disconnect between the two outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- AARDS Research, Inc, Aventura, Florida, United States

IPD SHARING:
Plan to Share IPD: No